CLINICAL TRIAL: NCT05822804
Title: Safety and Efficacy of the Vascular Closure Device (Tonbridge) in Hemostasis Treatment of Femoral Artery Puncture: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Trial
Brief Title: Safety and Efficacy of the Vascular Closure Device (Tonbridge) in Hemostasis Treatment of Femoral Artery Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ202204
Record Dates: First submitted 2023-04-05; First posted 2023-04-21 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-09

CONDITIONS: Vascular Closure; Endovascular Procedure; Hemostasis; Femoral Artery; Puncture
MeSH Terms: interventions — Vascular Closure Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Vascular Closure Device (Tonbridge)
  Interventions: Device: Vascular Closure Device (Tonbridge)
- control group (Active Comparator): EXOSEAL Vascular Closure Device (Codis Corporation)
  Interventions: Device: EXOSEAL Vascular Closure Device (Codis Corporation)

INTERVENTIONS:
Device: Vascular Closure Device (Tonbridge) — Hemostasis treatment for femoral artery puncture with Vascular Closure Device (Tonbridge).
  Arms: experimental group
Device: EXOSEAL Vascular Closure Device (Codis Corporation) — Hemostasis treatment for femoral artery puncture with EXOSEAL Vascular Closure Device (Codis Corporation).
  Arms: control group

SUMMARY:
The purpose of this study is to verify the safety and efficacy of the Vascular Closure Device (Tonbridge) in hemostasis treatment for femoral artery puncture.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized control, non-inferiority clinical trial carried out in 7 centers throughout China. 228 subjects with hemostasis of femoral artery puncture will be treated with the Vascular Closure Device (Tonbridge) or the EXOSEAL Vascular Closure Device (Codis Corporation). The primary objective of this study is to evaluate the safety and effectiveness of the vascular closure device in hemostasis treatment for femoral artery puncture.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80, male or non-pregnant female;
* Subjects undergoing unilateral femoral artery retrograde puncture for angiography or interventional procedure;
* Using guide sheath ≥5F to ≤8F, and length ≤12cm in angiography or interventional procedure;
* Subjects or their legal guardians voluntarily participate in this study, can complete follow-ups, and sign the informed consent form.

Exclusion Criteria:

* Ipsilateral common femoral artery occlusion or lumen diameter < 5mm;
* Inability to walk;
* Allergy to contrast media;
* Allergy to PGA or PEG; subjects with a history of common femoral artery surgery, percutaneous transluminal angioplasty (PTA), stent implantation, or vascular graft;
* Subjects with bleeding tendency, such as thrombocytopenia (platelet count <100×109/L), hemophilia, von willebrand diseases, pre-procedure INR >1.5, etc.;
* Subjects have taken anticoagulants for a long term before the procedure and have blood coagulation disorders;
* BMI >40kg/m^2;
* Subjects receive thrombolytic therapy (such as streptokinase, urokinase, t-PA) within≤24 hours before vascular closure;
* Local infections or skin infections of the investigational limb;
* Subjects with target femoral artery dissection or aneurysm within 30 days before intervention procedure;
* Subjects with puncture site have been punctured through the posterior wall of the femoral artery, or have been punctured several times (≥3 times), or have bleeding or hematoma on the femoral artery puncture site during the procedure;
* Subjects with clinically significant peripheral vascular diseases (such as severe calcification, arteritis, stenosis, etc) near the puncture site;
* Women who are pregnant or breastfeeding, OR men or women who plan to have a child in the next 6 months;
* Subjects who are enrolled in other clinical trials and don't complete;
* Subjects are considered not suitable for enrollment by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Immediate hemostasis success rate | intra-procedure
  Immediate hemostasis success is defined as no significant blood oozing and no visible or palpable expanding or developing hematoma on femoral artery puncture site within 5 minutes, once completing the closure operation of femoral artery puncture site using vascular closure device.

SECONDARY OUTCOMES:
Time to hemostasis | intra-procedure
  The time it takes (unit: minute) to reach no significant blood oozing and no visible or palpable expanding or developing hematoma on femoral artery puncture site, once completing the closure operation of femoral artery puncture site using vascular closure device.
Incidence of complications associated with femoral artery access | 30±7 days post-procedure
  "Incidence of complications associated with femoral artery access" is the proportion of subjects with femoral artery access complications using the investigational device or the comparator.
Incidence of device deficiency | intra-procedure
  Device deficiency is the unreasonable risk that may endanger human health and life safety under normal use of medical devices during clinical trials, such as labeling errors, quality problems and malfunctions, etc.
Incidence of adverse events (AE) | 30±7 days post-procedure
  "Incidence of adverse events" is the proportion of subjects with adverse events using the investigational device or the comparator.
Incidence of serious adverse events (SAE) | 30±7 days post-procedure
  "Incidence of serious adverse events" is the proportion of subjects with serious adverse events using the investigational device or the comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Tianxiao Li, Principal Investigator — Henan Provincial People's Hospital
Locations (7):
- China (7):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Nanyang Central Hospital, Nanyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No